CLINICAL TRIAL: NCT00314639
Title: The Impact of Modafinil as an Adjunctive to a Second Generation Antipsychotic on Cognitive Functioning in Schizophrenia and Schizophrenia Spectrum Psychosis.
Brief Title: Modafinil as an Adjunctive on Cognitive Functioning in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Dr Marc-André Roy, MD, FRCP, Centre de Recherche Université Laval Robert-Giffard
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4764
Record Dates: First submitted 2006-04-12; First posted 2006-04-14 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2007-04

CONDITIONS: Schizophrenia and Schizophrenia Spectrum Psychosis
MeSH Terms: conditions — Schizophrenia | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: modafinil — Modafinil OR Placebo 100mg orally (on the morning) from day 0 to day 14 and 200mg orally (on the morning) from day 15 to day 28. AND REVERSE : Modafinil OR Placebo 100mg orally (on the morning) from day 42 to day 56 and 200mg orally (on the morning) from day 57 to day 70.

SUMMARY:
Patients suffering from schizophrenia and schizophrenia spectrum psychosis frequently experience cognitive impairments. Such deficits may affect memory, attention and executive function processes. Many studies have shown that cognitive impairments predict daily functioning. Improvement of these difficulties represents a major component of recovery in such population. Second generation antipsychotics, now first line intervention, have been shown to improve cognitive processes compared to first generation agents. However, more subtle cognitive impairments may still remain. In fact, cognitive impairments is one of the most frequent subjective complaints from patients and their family, even though antipsychotic treatment has been optimized. Very few options are available to clinicians to try to improve such persistent cognitive difficulties. First, cognitive remediation techniques have shown some effectiveness but results are sparse and come from a very small number of studies. It is also not clear if cognitive improvement obtained from such techniques would apply to daily functioning and can be generalized.A second possible intervention would be to add a pharmacological agent able to improve cognition. Modafinil (Alertec) is officially indicated for improving wakefulness in patients with excessive daytime sleepiness associated with narcolepsy. Some empirical data and clinical observations suggest that modafinil could improve alertness and/or cognitive functioning without exacerbating psychotic features in persons with schizophrenia and psychotic disease in the spectrum of schizophrenia. This study aims to (a) assess the effect on cognitive functioning of modafinil as an adjunctive to a second generation antipsychotic in a prospective cohort of thirty patients suffering from schizophrenia and psychosis in the spectrum of schizophrenia. This study will also (b) evaluate the impacts of the addition of modafinil on side effects, psychopathology symptoms and other health parameters (such as weight, metabolic profile, etc.). Our principal hypothesis is that significant improvements will be observed on attention processes without any exacerbation of psychotic symptoms or major emerging side effects. This cross-over placebo-controlled prospective study will include patients with schizophrenia or psychosis in the schizophrenia spectrum according to DSM IV definition, men or women aged over 18 years old, with no item score equal or over 5 at PANSS positive symptoms subscale. At enrollment, all patients will have to experience significant cognitive difficulties with scores equal or lower than Z=-1.00 at Color trail test, Mesulam and Weintraub Cancellation Test, Stroop test or Continuous Performance Test-II. Patients will be exposed to 100mg daily of Placebo or Modafinil for 2 weeks than to 200mg daily for the two following weeks. A two weeks wash out period will then take place before the same sequence will be start again. Patient will thus be exposed one month to placebo and one month to modafinil or conversely, in a random fashion.Assessments will include neurocognitive standardized battery, psychopathological tools (PANSS, CGI, SOFAS, SDS), side effects (UKU, ESRS, DAI), vital signs, anthropometric and metabolic profile.

ELIGIBILITY:
Inclusion Criteria:

1. To have a diagnosis of schizophrenia or schizophrenia spectrum psychosis (schizophreniform, schizoaffective, delusional trouble, brief psychosis), as defined in Diagnostic and statistical manual of mental disorders ([DSM-IV], American Psychiatric Association [APA], 1995);
2. To be 18 years old or more;
3. Psychotic symptoms must be stabilized with a second generation antipsychotic for at least 4 weeks i.e. no item on Positive And Negative Syndrome Scale ([PANSS], Kay, Opler, & Fiszbein, 1987) positive subscale equal or superior to a score of 5.
4. Neurocognitive impairments are observed on attention measures. Participants will merit one or more result equal or lower to Z = -1,00 in at least one attention task.(Color trail test part A, MWCT, Stroop test, CPT-II).

Exclusion Criteria:

1. To have a diagnosis of mental retardation (APA, 1994), or medical affection other than schizophrenia or schizophrenia spectrum psychosis, or neurological troubles that can lead to cognitive impairments (ex : temporal epilepsy);
2. To have a current diagnosis of panic disorder (DSM-IV);
3. To manifest an important suicidal potential according to the psychiatrist clinical judgment;
4. To suffer from unstable hypertension, cardiac arrhythmia or any other cardiac disorders;
5. To take medications, drugs and/or natural products that have a stimulant effect on the CNS (e.g., cocaine, methylphenidate); and
6. To be a pregnant woman, who breast-feed, or a woman who do not use an effective contraceptive (abstinence is considered like an effective method).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-09; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Neuropsychological assessments | Pre and post Modafinil and Placebo Phases (Days 0, 28, 42 and 70)

SECONDARY OUTCOMES:
Psychiatric assessments | Pre, middle, & post Modafinil and Placebo phases (Days 0, 14, 28, 42, 56, 70)
Safety assessments | Pre, middle, & post Modafinil and Placebo phases (Days 0, 14, 28, 42, 56, 70)

CONTACTS AND LOCATIONS:
Overall Officials: Marc-André Roy, MD,MSc,FRCP, Principal Investigator — Centre de Recherche Université Laval Robert-Giffard
Locations (1):
- Centre Hospitalier Robert-Giffard, Québec, Quebec, Canada